CLINICAL TRIAL: NCT06948149
Title: Examining the Effects of Creatine Supplementation and Resistance Training on Cognition and Brain Health in Older Adults With Mild Cognitive Impairment: a 26 Week Randomized Controlled Trial
Brief Title: Creatine and Resistance Training in Older Adults With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Principal Investigator, Lindsay Nagamatsu, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: WesternUCanada1
Record Dates: First submitted 2024-10-10; First posted 2025-04-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Creatine; Exercise; Mild Cognitive Impairment (MCI)
Keywords: older adults; physical activity; cognition; neuroimaging; mobility; Mild Cognitive Impairment
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction | interventions — Creatine; Resistance Training

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a 26-week double blinded randomized controlled trial using a 2x2 factorial design, with factors of creatine supplementation (vs. placebo) and resistance training (vs. active control). Participants will be randomly assigned to one of the four groups.
  Sample size calculations in G*Power show that for an ANCOVA statistical analysis assuming a medium effect size (f = 0.25; np2 = 0.06) for the primary outcome measure, alpha=0.05, power=0.80, covariates=1 (baseline Corsi scores) a total sample size of 179 participants is required. Conservatively estimating ~10% drop out, a total of 200 participants (50 per group) will be recruited.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, physicians, and researchers who assess outcomes at endpoint will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Creatine monohydrate supplementation and resistance training (Experimental): Creatine supplementation: Participants will consume one serving (0.10g of creatine/kg/day) of creatine monohydrate mixed into at least eight ounces of a beverage of their choice daily. Participants will choose what meal they will take the supplement and will be asked to keep timing consistent throughout the 26 weeks.
  Resistance training: All participants will attend three 60-minute exercise classes per week. Classes will consist of a 10-minute warm-up on a treadmill or stationary bike followed up 40 minutes of core-content and ending with a 10-minute cool down and stretch. Resistance training classes will be completed using HUR machines which will target each major muscle group. Progression will follow the 7RM method where load will increase after two sets of 6-8 repetitions can be completed with proper form and range of motion.
  Interventions: Dietary Supplement: Creatine monohydrate; Behavioral: Resistance training
- Creatine monohydrate supplementation and active control group (Experimental): Creatine supplementation: Participants will consume one serving (0.10g of creatine/kg/day) of creatine monohydrate mixed into at least eight ounces of a beverage of their choice daily. Participants will choose what meal they will take the supplement and will be asked to keep timing consistent throughout the 26 weeks.
  Active control group: This group will follow the same protocol as the resistance training group, however, the core-content will consist of balance, stretching, and range of motion exercises. This serves as our active control group to control for socialization and commitment to an exercise program that may influence our outcome measures. This protocol has been used in previous exercise studies and there is no evidence that the balance and tone classes result in cognitive benefits.
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo supplementation and resistance training (Experimental): Placebo supplementation: Participants in the placebo group will follow the same protocol as the creatine supplementation groups but will consume dextrose powder instead of creatine.
  Resistance training: All participants will attend three 60-minute exercise classes per week. Classes will consist of a 10-minute warm-up on a treadmill or stationary bike followed up 40 minutes of core-content and ending with a 10-minute cool down and stretch. Resistance training classes will be completed using HUR machines which will target each major muscle group. Progression will follow the 7RM method where load will increase after two sets of 6-8 repetitions can be completed with proper form and range of motion.
  Interventions: Behavioral: Resistance training
- Placebo supplementation and active control group (No Intervention): Placebo supplementation: Participants in the placebo group will follow the same protocol as the creatine supplementation groups but will consume dextrose powder instead of creatine.
  Active control group: This group will follow the same protocol as the resistance training group, however, the core-content will consist of balance, stretching, and range of motion exercises. This serves as our active control group to control for socialization and commitment to an exercise program that may influence our outcome measures. This protocol has been used in previous exercise studies and there is no evidence that the balance and tone classes result in cognitive benefits.

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Participants will consume one serving of creatine daily (0.10g of creatine/kg of body weight). This relative dosing approach ensures that smaller participants do not receive excessive doses, while larger participants receive an adequate amount. There is currently limited evidence to conclude the effectiveness of timing daily creatine intake, but it is recommended that creatine be consumed at mealtime for optimal absorption. Participants will choose what meal they will take the supplement and will be asked to keep timing consistent throughout the study. This daily low dose method was chosen because other methods (high-dose loading) may have negative side effects (e.g., water retention, cramping).
  Arms: Creatine monohydrate supplementation and active control group; Creatine monohydrate supplementation and resistance training
Behavioral: Resistance training — Participants will use the programmable weight machines along with free weights to target primary muscle groups. In addition, they will complete mini-squats, mini-lunges, and lunge walks. Participants will complete two sets of 6-8 reps. Training stimulus will be increased using the 7RM method - when 2 sets of 6-8 reps are completed with proper form and without discomfort. The investigators will record the number of sets completed and the load lifted for each exercise for each participant at every class.
  Arms: Creatine monohydrate supplementation and resistance training; Placebo supplementation and resistance training

SUMMARY:
The goal of this 26-week trial is to learn if creatine supplementation and resistance training (i.e., weightlifting; exercise that increases muscle mass), alone and together, impact cognition, brain health, and physical function in older adults with mild cognitive impairment. Previous studies have shown that resistance training improves cognition and brain health in older adults. Creatine is naturally occurring in the human body and is known to decline with age. Studies have shown that creatine increases muscle mass and bone density in older adults when supplemented. Some research has suggested that creatine may also improve cognition and brain health. However, little is known about how creatine supplementation affects the aging brain and body alone and when combined with resistance training, especially in those with known cognitive impairment.

In this study, participants will be randomly assigned to one of four groups: 1) creatine and resistance training, 2) placebo and resistance training, 3) creatine and active control (balance and tone classes), or 4) placebo and active control. Participants in the creatine groups will take creatine every day during the study. Participants in the placebo groups will take a look-alike substance that contains no drug every day during the study. Participants in the resistance training groups will attend three 60-minute classes per week that target each major muscle group and will increase in difficulty during the study. Participants in the active control group will attend three 60-minute classes per week that will consist of balance, stretching, and range of motion exercises. This group accounts for variables such as physical training received by traveling to the training centres, social interaction, and changes in lifestyle secondary to study participation.

Researchers will collect information before and after the 26 weeks to see if creatine supplementation and/or resistance training have any effects on cognition, brain health, and/or physical function. The investigators suspect that both creatine supplementation and resistance training will improve cognition, brain health, and physical function alone. However, it is thought that the combination of creatine supplementation and resistance training will improve cognition, brain health, and physical function more.

DETAILED DESCRIPTION:
Research objectives:

To evaluate the effects of 26 weeks of creatine supplementation on its own and in combination with progressive resistance training in community-dwelling older adults with mild cognitive impairment on:

1. visuospatial working memory (Primary Objective);
2. executive function (working memory, inhibitory control, and mental flexibility), functional mobility, muscle and grip strength, bone density, cerebral blood flow, and blood-based biomarkers for brain health and cognitive decline (Secondary Objectives); and
3. resting state functional activity, hippocampal volume and structural integrity, and key metabolite concentrations in the brain (Exploratory Objective).

Hypotheses:

It is hypothesized that 26 weeks of creatine supplementation and resistance training in community-dwelling older adults with mild cognitive impairment will: 1) increase visuospatial working memory performance; 2) improve executive function, functional mobility, strength performance, bone density, cerebral blood flow, and blood-based biomarkers for brain health and cognitive decline; and 3) increase resting state functional activity, volume and structural integrity in the hippocampus, and concentrations of key metabolites in the brain.

Methods:

Screening: Participants interested in the study will reach out to researchers via phone or e-mail. Interested participants will be sent the Letter of Information via e-mail to get more detailed information about the study. Before a baseline assessment is scheduled, investigators will complete an initial screening over the phone with all participants to ensure that study eligibility is met. The Physical Activity Readiness Questionnaire (PAR-Q) will be administered over the phone as part of initial screening to ensure that they can partake in exercise. At this time, participants will have an opportunity to ask questions. Those who are eligible and still interested in participating will be scheduled to come into the lab for baseline assessments.

Baseline assessments: When participants arrive in the lab, the researcher will go over the consent form with them, answer any additional questions they have about the study, and obtain informed written consent. At this time, participants may also consent to participate in the optional MRI portion of this study. Participants will then complete baseline assessments. Total time to complete baseline assessments in the lab (excluding MRI) will be ~2.5-3 hours. For those participating in the MRI component, this will be scheduled for another separate visit (1 hour).

Randomization: Once participants complete baseline assessment, they will be randomly assigned to one of the four conditions. Group allocation will be determined by an online randomizer (randomization.com). The sequence will be held remotely by the PI and will not be revealed until after baseline assessments.

Descriptors and covariates:

1. Anthropometry (height, weight)
2. Demographic information via general questionnaire (e.g., age, sex, gender, ethnicity, education, socioeconomic status)
3. Global cognitive function (Montreal Cognitive Assessment, MoCA; Mini-Mental Status Examination, MMSE). MoCA is used as a screening tool for mild cognitive impairment. This test assesses cognitive ability in the domains of attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. Maximum score is 30. The MMSE is used as a screening tool for cognitive impairment. This 11-item test assesses global cognitive function in the domains of orientation, registration, attention and calculation, recall, and language. Maximum score is 30.
4. Physical activity levels (Physical Activities Scale for the Elderly, PASE). Used to measure the level of self-reported physical activity, and consists of 12 questions about leisure, household, and work-related daily activity.
5. Mood (Depression Scale, GDS).The GDS is a 15-item questionnaire used to test for the presence of depression. If depression is suspected, the PI will ensure that the participant is provided with a copy of the questionnaire and will advise the participant to make an appointment with their family physician to discuss the results.
6. Number of co-morbidities (Functional Comorbidity Index, FCI). The FCI is an 18-item list of diagnoses used to determine co-morbidities.
7. Health-related quality of life (Short Form Health Survey, SF-12). A self-reported questionnaire that measures a person's health-related quality of life and functional health status. Developed as a shorter alternative to the original SF-36 survey, the SF-23 assesses eight different health domains (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health) and provides summary scores for physical and mental health. Scores range from 0-100, with higher scores indicating greater health status and quality of life.
8. Loneliness (UCLA, Loneliness Scale). A 20-item self report measure on loneliness and interpersonal problems.

Adherence: All participants will be asked to record their supplement consumption on a calendar, which will be returned to the lab weekly. Exercise class attendance will be recorded each session by instructors. Participants will be encouraged to adhere to both the supplement protocol and exercise classes. The investigators will implement the following strategies to promote participant engagement:

* Semi-monthly newsletters that will feature personal accomplishments of participants (with permission) and study updates, for example.
* Investigators will follow up with participants who have missed supplement doses or exercise sessions to discuss barriers and strategies to overcome them on an individual basis.

If participants miss classes due to illness/travel, they will be scheduled to make up missing classes as soon as possible. If participants miss classes without notifying investigators in advance, investigators will call to remind them about their classes and encourage increased compliance.

During the 26-week intervention, participants will also complete the following assessments:

1. PASE (described in baseline assessments) - This will be used to monitor exercise outside of the program and will be administered at the last exercise session of each month.
2. Falls - Because declines in mobility are known to co-occur with declines in cognition, the investigators will monitor falls throughout the study duration to further characterize our sample. Participants will be asked to note falls in their calendar if they occur, which as mentioned above will be returned to the lab weekly for review by instructors.
3. Dietary intake - A three day weighed food record will be used to assess nutrient and energy intake at baseline and endpoint. Participants will record their dietary consumption over three days per month (two weekday and one weekend day). They will be instructed on how to do the food record at the first exercise session and will be asked to return it by the last exercise session of that month. The endpoint food record will be given to participants at the first session of the last month of the intervention and they will be asked to return it by the last exercise session of the month. A dietetic student will assist in analyzing this data.
4. Real-time physical activity levels will be monitored using wearable accelerometers (ActiGraph ambulatory monitoring wearables). Participants will be given the accelerometer to wear on their wrist for at baseline (one week during the first month of the intervention) and endpoint (one week during the last month of the intervention). This will allow objective quantification of energy expenditure, metabolic equivalent of task rates, steps, physical activity intensity, sedentary bouts, and sleep latency. They are Bluetooth enabled for real-time data uploads and include a wear-time sensor to assess compliance.

Final assessment: All baseline assessments will be completed at endpoint (26 weeks). The sub-set of participants at baseline who underwent MRI will also undergo the MRI protocol at endpoint.

Data analysis: Behavioural data (cognitive assessments, mobility, and physical measures) will be analyzed in SPSS. Primary and secondary outcome measures will be examined using a two-way ANCOVA to examine main effects of creatine supplementation and resistance training as well as the interaction between the two factors. The investigators will use the intention to treat principle where all randomized participants will be included in the final analysis regardless of adherence to the intervention. MRI data will be analyzed in Freesurfer and FSL. MRI/MRS data will be analyzed in collaboration with an expert who is familiar with processing this data. Investigators will examine changes over the intervention and compare these changes between groups.

Significance of research: This research is the first to address a critical gap in the literature by examining the effects of creatine and resistance training alone and in conjunction on various measures of physical function, cognitive function, and brain health in older adults with MCI. In the context of an aging population and given the overall safety and accessibility of creatine and resistance training, the findings from our study may inform biomarker-driven, non-pharmalogical strategies and interventions to offset or defer further cognitive decline in older adults with MCI.

ELIGIBILITY:
To be eligible to participate in this study participants must:

1. be 60 years of age or older,
2. live independently in the community,
3. have normal or corrected-to-normal vision and hearing,
4. read, write, and speak English fluently,
5. be right-handed,
6. have subjective feelings of memory decline in the past 5 years,
7. have MoCA scores 19-25/30 (assessed at baseline session),
8. be able to exercise at a moderate pace using resistance training for 60 minutes 3x/week,
9. receive clearance from a physician to participate in an exercise program, and 10) receive confirmation from a physician that they meet all criteria to be included in this study.

Participants are ineligible if they:

1. cannot partake or commit to exercise training 3x/week for 26 weeks or have regularly (>1x/week) engaged in exercise training over the past 3 months;
2. cannot partake or commit to consuming a daily supplement for 26 weeks or consumed nutritional supplements containing creatine monohydrate over the past 3 months;
3. have a known allergy to creatine monohydrate or dextrose;
4. have been diagnosed with a neurological disorder (e.g., Alzheimer's disease, Parkinson's disease);
5. have pre-existing kidney disease, heart disease, or liver abnormalities;
6. have one or more uncontrolled chronic or psychiatric conditions (e.g., hypertension, diabetes, depression, anxiety);
7. are taking medication that may impact kidney function (e.g., non-steroidal anti-inflammatory drugs, such as ibuprofen and naproxen); or
8. are ineligible or uncomfortable with MRI (have metal or electronic implants, claustrophobia) or blood sampling.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Corsi Span - Corsi Block Tapping Task | Baseline and 26 weeks
  Visuospatial working memory will be assessed using the forward and reverse Corsi block-tapping task. Participants will be given an iPad to complete the task. In this task, participants will see nine BLUE blocks on the screen. For each trial, a sequence of blocks will turn RED one by one. Their task is to remember the order in which the blocks light up and then repeat the sequence in the same order (forward Corsi) or backwards (reverse Corsi) by tapping on the blocks. Participants will first complete two practice trials before the true trials to ensure that the instructions are understood. Sequences will become increasingly more difficult with a maximum sequence of nine and a minimum of 2. The maximum sequence number that each participant correctly reproduces (Corsi span) will be measured, where higher scores indicate better visuospatial working memory.
Reaction Time - Corsi Block Tapping Task | Baseline and 26 weeks
  Visuospatial working memory will be assessed using the forward and reverse Corsi block-tapping task. Participants will be given an iPad to complete the task. In this task, participants will see nine BLUE blocks on the screen. For each trial, a sequence of blocks will turn RED one by one. Their task is to remember the order in which the blocks light up and then repeat the sequence in the same order (forward Corsi) or backwards (reverse Corsi) by tapping on the blocks. Participants will first complete two practice trials before the true trials to ensure that the instructions are understood. Sequences will become increasingly more difficult with a maximum sequence of nine and a minimum of 2. Reaction time, or how fast the participant can reproduce each sequence, will be measured.

SECONDARY OUTCOMES:
Interference Score - Stroop Task | Baseline and 26 weeks
  Investigators will examine the interference score for each participant using the Stroop task. Participants are required to read the colour of the ink that each word is printed in and inhibit what the word actually says. The time to complete this test is recorded in seconds. Higher scores reflect better performance and less interference.
Span Capacity - Digits Forward and Backward Subtests | Baseline and 26 weeks
  Working memory using the Digits Forward and Backward subtests. Participants are required to memorize and recall a series of number lists both forward and backward. Span capacity (the largest sequence to be recalled) will be measured. The minimum sequence for the forward test is three and the maximum is nine. The minimum sequence for the backward test is two and the maximum is eight. Higher sequences reproduced indicate better working memory.
Time - Trail Making Test (Part B) | Baseline and 26 weeks
  Mental flexibility using the Trail Making Test (Part B). Participants will have to alternate between numbers and letters without removing the pen from the page. The time to complete this test is recorded in seconds.
Time - Timed Up & Go (TUG) Test | Baseline and 26 weeks
  A test of functional mobility. Participants are seated in a chair and must stand up, walk three meters at their usual pace, turn around, return to their chair, and sit back down. The time to complete each of two separate trials is recorded in seconds. Time will be averaged between the two trials.
Short Physical Performance Battery (SPPB) Score | Baseline and 26 weeks
  Used to assess gait speed, balance, and lower extremity physical function using tasks that mimic daily activities; includes three tasks: 1. Standing Balance Task: participants stand unassisted (side-by-side standing, semi-tandem standing, and tandem standing) for a period of 10 seconds each; 2. Walking Speed Task: participants walk 4 metres at their usual pace; and 3. Chair Stand Test: participants stand up from a chair 5 times consecutively (without the use of their arms if possible). For task 1, participants receive the point(s) if they can hold the balance task for at least 10 seconds. Time to complete tasks 2 and 3 is recorded in seconds. The task is scored out of 12, with higher scores indicating better physical performance.
Falls History Questionnaire | Baseline and 26 weeks
  General questionnaire used to assess mobility and falls risk. The questionnaire asks the participant if they have fallen in the past six months. If no, the questionnaire is complete. If yes, participants continue to answer questions about the fall(s) (e.g., number of falls, any injuries, who witnessed the fall).
One Repetition Maximum (1RM) - Muscle Strength | Baseline and 26 weeks
  Muscle strength measured by 1RM testing. 1RM is a physical measure of an individual's maximum muscle strength during a single repetition and is used to determine the desired load for resistance training. Exercise includes leg press, latissimus pulldown, leg curl, chest press, bicep curls, tricep extensions, and pulley rows. 1RM testing will be performed at the first exercise session for each participant.
Grip Strength | Baseline and 26 weeks
  Measured using a calibrated hand dynamometer. Participants will be instructed to sit with their elbow at 90 degrees, wrist in a neutral position, and squeeze the dynamometer with maximal effort for 3-5 seconds. Three trials will be performed and recorded per hand, with 30 seconds of rest between attempts.
Bone Density | Baseline and 26 weeks
  Observed via dual-energy x-ray absorptiometry (DEXA or DXA). This is a common, non-invasive method often used to identify osteoporosis and fracture risk in older adults. Participants lay still on a padded table and an x-ray is taken of their entire body.
Muscle Mass | Baseline and 26 weeks
  Observed via dual-energy x-ray absorptiometry (DEXA or DXA). Participants lay still on a padded table and an x-ray is taken of their entire body.
Cerebral Blood Flow Velocity | Baseline and 26 weeks
  Measured using a transcranial doppler ultrasound (TCD). The TCD probe will be covered with ultrasound gel, placed on the left temple, and stabilized using a headband. The TCD emits ultrasound waves that provide a measure of cerebral blood velocity. TCD is safe, non-invasive and has been used extensively in previous work without any reported adverse effects.
Biomarker Concentration - Phosphorylated Tau 217 (p tau 217) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Higher levels of p tau 217 biomarker in blood plasma may suggest cognitive decline and progression to Alzheimer's disease.
Biomarker Concentration - Neurofilament Light Chain (NfL) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Higher plasma NfL levels are associated with cognitive decline.
Biomarker Concentration - Glial Fibrillary Acidic Protein (GFAP) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Elevated GFAP plasma levels have been shown to be elevated in those with cognitive decline.
Biomarker Concentration - Amyloid Beta 42 (Aβ42) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Low levels of Aβ42 in plasma have been linked to cognitive decline.
Biomarker Concentration - Creatinine | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Creatinine is a waste product formed from creatine breakdown. Creatinine levels in blood plasma should be elevated with creatine supplementation.
Biomarker Concentration - Brain-Derived Neurotrophic Factor (BDNF) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. BDNF is important for neuronal growth and plasticity. Some studies suggest that BDNF plasma levels may be lower in individuals with cognitive decline.
Biomarker Concentration - Insulin-like Growth Factor 1 (IGF-1) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. IGF-1 promotes neuronal growth and better cognitive function. Lower IGF-1 plasma levels are associated with cognitive decline.
Biomarker Concentration - Interleukin 6 (IL-6) | Baseline and 26 weeks
  Measured from blood samples and examined using a blood assay kit. Elevated IL-6 levels in blood plasma are associated with poorer cognitive performance and an increased risk of cognitive decline.
Six Minute Walk Test | Baseline and 26 Weeks
  Used as a proxy to assess cardiorespiratory fitness. The distance walked in six minutes is recorded.

OTHER OUTCOMES:
Hippocampal Volume - Structural MRI | Baseline and 26 weeks
  Hippocampal volume will be examined in a sub-set of participants using MRI. Participants will undergo structural MRI on the 3T Siemens scanner at the Centre for Functional and Metabolic Mapping (CFMM) on Western University campus. Participants will complete T1 and T2 high resolution anatomical scans.
Structural Integrity - Structural MRI | Baseline and 26 weeks
  Structural integrity will be examined in a sub-set of participants using MRI. Participants will undergo diffusion tensor imaging (DTI) on the 3T Siemens scanner at the Centre for Functional and Metabolic Mapping (CFMM) on campus. DTI allows for evaluation of microstructures in the brain by measuring water movement.
Resting State Functional Connectivity - Functional MRI | Baseline and 26 weeks
  Participants will be asked to remain as still as possible with eyes open while a 12-minute functional scan is performed. This will allow the investigators to examine activation in the resting state network.
Magnetic Resonance Spectroscopy - Functional MRI | Baseline and 26 weeks
  Provides information on metabolic activity in the brain. This technique will be used to examine key concentrations in the brain relevant to our study (e.g., creatine).

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vandierendonck A, Kemps E, Fastame MC, Szmalec A. Working memory components of the Corsi blocks task. Br J Psychol. 2004 Feb;95(Pt 1):57-79. doi: 10.1348/000712604322779460. PMID 15005868
- [Background] Swanson HL. Verbal and visual-spatial working memory: What develops over a life span? Dev Psychol. 2017 May;53(5):971-995. doi: 10.1037/dev0000291. PMID 28459277
- [Background] McMorris T, Mielcarz G, Harris RC, Swain JP, Howard A. Creatine supplementation and cognitive performance in elderly individuals. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2007 Sep;14(5):517-28. doi: 10.1080/13825580600788100. PMID 17828627
- [Background] Alves CR, Santiago BM, Lima FR, Otaduy MC, Calich AL, Tritto AC, de Sa Pinto AL, Roschel H, Leite CC, Benatti FB, Bonfa E, Gualano B. Creatine supplementation in fibromyalgia: a randomized, double-blind, placebo-controlled trial. Arthritis Care Res (Hoboken). 2013 Sep;65(9):1449-59. doi: 10.1002/acr.22020. PMID 23554283
- [Background] Forbes SC, Candow DG, Ferreira LHB, Souza-Junior TP. Effects of Creatine Supplementation on Properties of Muscle, Bone, and Brain Function in Older Adults: A Narrative Review. J Diet Suppl. 2022;19(3):318-335. doi: 10.1080/19390211.2021.1877232. Epub 2021 Jan 27. PMID 33502271
- [Background] Candow DG, Forbes SC, Chilibeck PD, Cornish SM, Antonio J, Kreider RB. Effectiveness of Creatine Supplementation on Aging Muscle and Bone: Focus on Falls Prevention and Inflammation. J Clin Med. 2019 Apr 11;8(4):488. doi: 10.3390/jcm8040488. PMID 30978926
- [Background] Xu L, Gu H, Cai X, Zhang Y, Hou X, Yu J, Sun T. The Effects of Exercise for Cognitive Function in Older Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2023 Jan 7;20(2):1088. doi: 10.3390/ijerph20021088. PMID 36673844
- [Background] Herold F, Torpel A, Schega L, Muller NG. Functional and/or structural brain changes in response to resistance exercises and resistance training lead to cognitive improvements - a systematic review. Eur Rev Aging Phys Act. 2019 Jul 10;16:10. doi: 10.1186/s11556-019-0217-2. eCollection 2019. PMID 31333805